CLINICAL TRIAL: NCT00288080
Title: A Phase III Protocol of Androgen Suppression (AS) and 3DCRT/IMRT Vs AS and 3DCTR/IMRT Followed by Chemotherapy With Docetaxel and Prednisone for Localized, High-Risk, Prostate Cancer
Brief Title: Hormone Therapy and Radiation Therapy or Hormone Therapy and Radiation Therapy Followed by Docetaxel and Prednisone in Treating Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0521; CDR0000462375; NCI-2009-00728 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer
Keywords: stage III prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dexamethasone; Prednisone; Docetaxel; Androgen Antagonists; Radiotherapy; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Androgen suppression + Radiation Therapy (Active Comparator): Androgen suppression (AS; LHRH agonist and oral antiandrogen) for 8 weeks followed by radiation therapy and concurrent AS. LHRH continues for 24 months after initiation of any treatment, oral antiandrogen discontinues at the end of radiation therapy (RT).
  Interventions: Drug: Oral antiandrogen; Radiation: Radiation therapy; Drug: LHRH agonist
- Androgen suppression + Radiation Therapy + Chemotherapy (Experimental): Androgen suppression (AS; LHRH agonist and oral antiandrogen) for 8 weeks followed by radiation therapy and concurrent AS. LHRH continues for 24 months after initiation of any treatment, oral antiandrogen discontinues at the end of RT. Following completion of RT, 6 cycles of docetaxel (premedicated with dexamethasone) and prednisone are delivered concurrently with androgen suppression.
  Interventions: Drug: Dexamethasone; Drug: Prednisone; Drug: docetaxel; Drug: Oral antiandrogen; Radiation: Radiation therapy; Drug: LHRH agonist

INTERVENTIONS:
Drug: Dexamethasone — Premedication of dexamethasone prior to docetaxel, per institutional standards.
  Arms: Androgen suppression + Radiation Therapy + Chemotherapy
Drug: Prednisone — 10 mg orally per day until day 21 of the last cycle of docetaxel, beginning 28 days after the completion of RT.
  Arms: Androgen suppression + Radiation Therapy + Chemotherapy
Drug: docetaxel — 75 mg/m2 i.v. over 1 hour (on day 1 of each cycle) every 21 days for 6 cycles, beginning 28 days after the completion of RT.
  Arms: Androgen suppression + Radiation Therapy + Chemotherapy
Drug: Oral antiandrogen — Oral antiandrogen of treating institution's choice to be given per package instructions for 8 weeks, then concurrent with radiation therapy. Treatment is discontinued at the end of radiation therapy.
Radiation: Radiation therapy — 46.8 Gy, using either three-dimensional conformal radiotherapy (3DCRT) or intensity-modulated radiation therapy (IMRT), will be given to the regional lymphatics followed by a 25.2-28.8 Gy boost to the prostate, to bring the total dose to the prostate to 72.0-75.6 Gy. Daily prescription doses will be 1.8 Gy per day, 5 days per week x 8-8.5 weeks, beginning 8 weeks after the initiation of androgen suppression.
  Other Names: 3DCRT; Three-dimensional conformal radiotherapy; IMRT; Intensity-modulated radiation therapy
Drug: LHRH agonist — LHRH agonist of treating institution's choice to be given per package instructions for 8 weeks, then concurrent with radiation therapy, and then until 24 months from initiation of any treatment has been reached.

SUMMARY:
RATIONALE: Androgens can cause the growth of prostate cancer cells. Hormone therapy using drugs, such as leuprolide, goserelin, flutamide, or bicalutamide, may fight prostate cancer by lowering the amount of androgens the body makes. Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as docetaxel and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving hormone therapy and radiation therapy together with chemotherapy is more effective than giving hormone therapy together with radiation therapy in treating prostate cancer.

PURPOSE: This randomized phase III trial is studying hormone therapy and radiation therapy followed by docetaxel and prednisone to see how well it works compared to hormone therapy and radiation therapy in treating patients with localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the relative efficacy, in terms of overall survival, of the combination of androgen suppression and radiotherapy versus androgen suppression and radiotherapy followed by docetaxel and prednisone in patients with localized, high-risk prostate cancer.

Secondary

* Compare the disease-free survival and incidence of adverse events in patients treated with these regimens.
* Compare the biochemical control, local control, and freedom from distant metastases in patients treated with these regimens.
* Determine the validity of prostate-specific antigen (PSA)-defined endpoints as a surrogate for overall survival of patients treated with these regimens.
* Compare the time interval between biochemical failure and distant metastases with respect to testosterone level in patients treated with these regimens.

OUTLINE: This is an open-label, randomized, multicenter study. Patients are stratified according to risk group.

* Arm I: Patients receive androgen suppression therapy comprising luteinizing hormone-releasing hormone (LHRH) agonist (e.g., leuprolide acetate, goserelin, buserelin, or triptorelin) and oral antiandrogen (i.e., oral flutamide 3 times daily for 2 months or oral bicalutamide once daily for 2 months). Beginning at week 8, patients undergo radiotherapy 5 days a week for approximately 8 weeks. Antiandrogen therapy is discontinued at completion of radiotherapy, but LHRH agonist therapy continues for 20 months.
* Arm II: Patients receive androgen suppression therapy and undergo radiotherapy as in arm I. Beginning 4 weeks after completion of radiotherapy, patients receive docetaxel IV over 1 hour on day 1 and oral prednisone daily on days 1-21. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients continue LHRH agonist therapy as in arm I.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 600 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed prostate cancer at high-risk for recurrence within the past 180 days as determined by 1 of the following combinations (risk groups):

  * Gleason score ≥ 9, prostate-specific antigen (PSA) ≤ 150 ng/mL, and any T stage
  * Gleason score 8, PSA < 20 ng/mL, and stage ≥ T2
  * Gleason score 8, PSA 20-150 ng/mL, and any T stage
  * Gleason score 7, PSA 20-150 ng/mL, and any T stage
* Clinically negative lymph nodes by imaging (pelvic CT scan or pelvic MRI), nodal sampling, or dissection within 90 days prior to study entry

  * Equivocal or questionable lymph nodes ≤ 1.5 cm by imaging allowed
  * Positive lymph nodes by capromab pendetide (ProstaScint^®) scan with a corresponding lymph node ≤ 1.5 cm by CT scan or MRI allowed
* PSA ≤ 150 ng/mL

  * Cannot have been obtained during any of the following time points:

    * 10-day period after prostate biopsy
    * After initiation of hormonal therapy
    * Within 30 days after discontinuation of finasteride
    * Within 90 days after discontinuation of dutasteride
* No distant metastases by physical exam and bone scan

  * Equivocal bone scan findings allowed if plain films are negative

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count ≥ 1,800/mm^3
* Hemoglobin ≥ 8 g/dL (transfusion or other intervention allowed)
* Alanine transaminase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Bilirubin ≤ 1.5 times ULN
* Fertile patients must use effective contraception during and for at least 3 months after completion of study treatment
* No prior invasive malignancy, except nonmelanomatous skin cancer or other malignancy, unless disease-free for ≥ 3 years (e.g., carcinoma in situ of the oral cavity or bladder are allowed)
* No unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
* No transmural myocardial infarction within the past 6 months
* No acute bacterial or fungal infection requiring intravenous antibiotics
* No AIDS
* No prior allergic reaction to any study drugs or other drugs formulated with polysorbate 80
* No existing peripheral neuropathy ≥ grade 2

PRIOR CONCURRENT THERAPY:

* At least 60 days since prior 5-alpha reductase inhibitor (e.g., finasteride) for prostatic hypertrophy
* At least 90 days since prior testosterone
* Prior pharmacologic androgen ablation for prostate cancer allowed provided androgen ablation was initiated no more than 50 days prior to study entry
* No prior radical prostatectomy, cryosurgery for prostate cancer, or bilateral orchiectomy
* No prior systemic chemotherapy for prostate cancer

  * Prior chemotherapy for a different cancer is allowed
* No prior radiotherapy, including brachytherapy, to the region of prostate cancer that would result in overlap of radiotherapy fields
* Intensity modulated radiotherapy allowed

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2005-12; Primary Completion 2014-04 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard M. Sandler, MD, Principal Investigator — University of Michigan Rogel Cancer Center; Seth Rosenthal, MD, Study Chair — Radiological Associates of Sacramento Medical Group at Sutter Cancer Center; Mahul Amin, MD, Study Chair — Cedars-Sinai Medical Center; Leonard G. Gomella, MD, Study Chair — Sidney Kimmel Cancer Center at Thomas Jefferson University; James Purdy, PhD, Study Chair — University of California, Davis; Jeff Michalski, MD, Study Chair — Washington University School of Medicine; Mark Garzotto, MD, Study Chair — Portland VA Medical Center; Oliver Sartor, MD, Study Chair — Tulane School of Medicine
Locations (254):
- United States (245):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Providence Cancer Center, Anchorage, Alaska
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Arizona Oncology - Tucson, Tucson, Arizona
  - Auburn Radiation Oncology, Auburn, California
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - Enloe Cancer Center at Enloe Medical Center, Chico, California
  - Cancer Care Center at John Muir Health - Concord Campus, Concord, California
  - Washington Township Hospital, Fremont, California
  - Sierra Nevada Cancer Center at Sierra Nevada Memorial Hospital, Grass Valley, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Memorial Medical Center, Modesto, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Lucy Curci Cancer Center at Eisenhower Memorial Hospital and Medical Center, Rancho Mirage, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Torrance Memorial Medical Center, Torrance, California
  - Solano Radiation Oncology Center, Vacaville, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Radiation Oncology, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - St. Vincent's Medical Center, Bridgeport, Connecticut
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Hospital of Saint Raphael, New Haven, Connecticut
  - Yale Cancer Center, New Haven, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - William W. Backus Hospital, Norwich, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Bay Medical, Panama City, Florida
  - Georgia Cancer Center for Excellence at Grady Memorial Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Center for Cancer Care at OSF Saint Anthony Medical Center, Rockford, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Saint John's Cancer Center at Saint John's Medical Center, Anderson, Indiana
  - Radiation Oncology Associates Southwest, Fort Wayne, Indiana
  - Parkview Regional Cancer Center at Parkview Health, Fort Wayne, Indiana
  - Veterans Affairs Medical Center - Indianapolis, Indianapolis, Indiana
  - Central Indiana Cancer Centers - East, Indianapolis, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Kansas City Cancer Centers - Southwest, Overland Park, Kansas
  - Norton Suburban Hospital, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Center for Cancer Medicine and Blood Disorders - Scarborough, Scarborough, Maine
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Shields Radiation Oncology Center - Mansfield, Mansfield, Massachusetts
  - NSMC Cancer Center - Peabody, Peabody, Massachusetts
  - South Suburban Oncology Center, Quincy, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Cancer Institute of Cape Girardeau, LLC, Cape Girardeau, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - Kansas City Cancer Centers - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Dartmouth - Hitchcock Concord, Concord, New Hampshire
  - Seacoast Cancer Center at Wentworth - Douglass Hospital, Dover, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Cancer Institute of New Jersey at Cooper University Hospital - Camden, Camden, New Jersey
  - CentraState Medical Center, Freehold, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - Radiation Oncology Associates, PA, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Cancer Institute of New Mexico, Santa Fe, New Mexico
  - New York Oncology Hematology, PC at Albany Regional Cancer Care, Albany, New York
  - Bassett Healthcare Regional Cancer Program at Mary Imogene Bassett Hospital, Cooperstown, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CaroMont Cancer Center at Gaston Memorial Hospital, Gastonia, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - New Hanover Radiation Oncology, PA, Wilmington, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Willamette Valley Cancer Center - Eugene, Eugene, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Celilo Cancer Center at Mid-Columbia Medical Center, The Dalles, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - UPMC Cancer Center at Beaver Medical Center, Beaver, Pennsylvania
  - UPMC Cancer Center at Jefferson Regional Medical Center, Clairton, Pennsylvania
  - Cancer Center at Clarion Hospital, Clarion, Pennsylvania
  - Mercy Fitzgerald Hospital, Darby, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - UPMC Cancer Center - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Cancer Center at the John P. Murtha Pavilion, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC - Moon, Moon Township, Pennsylvania
  - UPMC Cancer Center - Natrona Heights, Natrona Heights, Pennsylvania
  - Jameson Memorial Hospital - North Campus, New Castle, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - UPMC - Shadyside, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC St. Margaret, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Passavant, Pittsburgh, Pennsylvania
  - UPMC Cancer Center - Upper St. Clair, Pittsburgh, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center - Uniontown, Uniontown, Pennsylvania
  - Washington Hospital Cancer Center, Washington, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Texas Oncology, PA at Harris Center HEB, Bedford, Texas
  - St. Joseph Regional Cancer Center, Bryan, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Texas Oncology, PA at Texas Cancer Center Dallas Southwest, Dallas, Texas
  - Klabzuba Cancer Center at Harris Methodist Fort Worth Hospital, Fort Worth, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Texas Oncology, PA at Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology, PA at Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Community Cancer Center at Rutland Regional Medical Center, Rutland, Vermont
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Theda Care Cancer Institute, Appleton, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Community Memorial Hospital Cancer Care Center, Menomonee Falls, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia-Saint Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
- Canada (9):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan

REFERENCES:
- [Result] Patel AR, Sandler HM, Pienta KJ. Radiation Therapy Oncology Group 0521: a phase III randomized trial of androgen suppression and radiation therapy versus androgen suppression and radiation therapy followed by chemotherapy with docetaxel/prednisone for localized, high-risk prostate cancer. Clin Genitourin Cancer. 2005 Dec;4(3):212-4. doi: 10.3816/cgc.2005.n.035. No abstract available. PMID 16425991
- [Derived] Phillips RM, Proudfoot JA, Davicioni E, Liu Y, Spratt DE, Simko JM, Den RB, Pollack A, Rosenthal SA, Sartor AO, Sweeney CJ, Attard G, Longoria L, Patel S, Straza MW, Efstathiou JA, Shah AB, Hoffman KE, Rodgers JP, Sandler HM, Feng FY, Tran PT. Transcriptomic Analysis of Localized High-risk Prostate Cancer Improves Prognostication and Identifies Benefit from Adding Docetaxel to Definitive Radiotherapy with Androgen Suppression in the NRG Oncology/RTOG 0521 Phase 3 Trial. Eur Urol Oncol. 2025 Aug;8(4):968-976. doi: 10.1016/j.euo.2025.04.009. Epub 2025 Jul 17. PMID 40675873
- [Derived] Flannery BT, Sandler HM, Lal P, Feldman MD, Santa-Rosario JC, Pathak T, Mirtti T, Farre X, Correa R, Chafe S, Shah A, Efstathiou JA, Hoffman K, Hallman MA, Straza M, Jordan R, Pugh SL, Feng F, Madabhushi A. Stress testing deep learning models for prostate cancer detection on biopsies and surgical specimens. J Pathol. 2025 Feb;265(2):146-157. doi: 10.1002/path.6373. Epub 2024 Dec 11. PMID 39660731
- Available data/document: Individual Participant Data Set: NCT00288080 — https://nctn-data-archive.nci.nih.gov/ — Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

RESULTS

PARTICIPANT FLOW:
Groups:
- Androgen Suppression + Radiation Therapy (RT): Androgen suppression (AS; luteinizing hormone-releasing hormone (LHRH) agonist and oral antiandrogen) for 8 weeks followed by radiation therapy and concurrent AS. LHRH continues for 24 months after initiation of any treatment, oral antiandrogen discontinues at the end of RT.
Period: Overall Study
Arm/Group | Androgen Suppression + Radiation Therapy (RT) | Androgen Suppression + Radiation Therapy + Chemotherapy
Started | 307 | 305
Completed | 281 (Subjects with data available for the primary analysis are considered to have completed the study.) | 282 (Subjects with data available for the primary analysis are considered to have completed the study.)
Not Completed | 26 | 23
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 25 | 20

BASELINE CHARACTERISTICS:
Population: Eligible patients who have not withdrawn consent.
Groups:
- Androgen Suppression + Radiation Therapy: Androgen suppression (AS; LHRH agonist and oral antiandrogen) for 8 weeks followed by radiation therapy and concurrent AS. LHRH continues for 24 months after initiation of any treatment, oral antiandrogen discontinues at the end of RT.
- Total: Total of all reporting groups
Arm/Group | Androgen Suppression + Radiation Therapy | Androgen Suppression + Radiation Therapy + Chemotherapy | Total
Number analyzed (Participants) | 281 | 282 | 563
Age, Continuous [Median (Full Range); unit: years] | 66 [47 to 83] | 66 [46 to 83] | 66 [46 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 281 | 282 | 563

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Four-year rates are shown. Survival time is defined as time from randomization to date of death from any cause and is estimated by the Kaplan-Meier method. Patients last known to be alive are censored at the date of last contact.
Time Frame: From randomization to date of death or last follow-up. Analysis occurs after all patients have been potentially followed for 4 years.
Population: Eligible patients who did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Androgen Suppression + Radiation Therapy | Androgen Suppression + Radiation Therapy + Chemotherapy
Number analyzed (Participants) | 281 | 282
percentage of participants | 88.7 [84.3 to 91.9] | 93.3 [89.6 to 95.7]
Statistical Analysis 1: Comparison: Androgen Suppression + Radiation Therapy vs Androgen Suppression + Radiation Therapy + Chemotherapy; The study was designed to detect an improvement in the 4-year overall survival rate from 86% (AS+RT) to 93% (AS+RT+CT). Assuming an exponential survival distribution for each arm, then an absolute improvement of 7% in the 4-year overall survival rate translates to a 51% relative reduction (hazard ratio 0.49) in the yearly death rate. Under a 1-sided significance level of 0.05 and 90% power, at least 78 deaths and 486 cases were required to perform the primary endpoint analysis; Test type: Superiority or Other; p = 0.0398, Log Rank

2. Secondary Outcome: Biochemical Control
Description: Four-year rates are shown (Kaplan-Meier estimates). Biochemical control is defined as freedom from biochemical failure. Biochemical failure was considered as the first of either prostate-specific antigen (PSA) failure or initiation of salvage hormone therapy. PSA failure was defined as a rise of 2 ng/ml over the nadir PSA. Patients who experienced death without biochemical failure, local failure prior to biochemical failure, or development of distant metastases prior to biochemical failure were censored on the date of the competing event. The corresponding outcome time was measured from the date of randomization.
Time Frame: From randomization to date of biochemical failure, death, or last follow-up. Analysis occurs after all patients have been potentially followed for 4 years.
Population: Eligible patients who did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Androgen Suppression + Radiation Therapy | Androgen Suppression + Radiation Therapy + Chemotherapy
Number analyzed (Participants) | 281 | 282
percentage of participants | 82.0 [76.7 to 86.1] | 84.1 [79 to 88]
Statistical Analysis 1: Comparison: Androgen Suppression + Radiation Therapy vs Androgen Suppression + Radiation Therapy + Chemotherapy; Biochemical control rates at 4 years were calculated using the Kaplan-Meier method and compared by a two-sided log-rank test with a significance level of 0.05; Test type: Superiority or Other; p = 0.22, Log Rank

3. Secondary Outcome: Local Control
Description: Local control is defined as the absence of local failure which is the first of either progression or recurrence within the prostate. Progression of the tumor was considered to have occurred when there was a 25% or greater increase in the product of the two largest perpendicular diameters of the prostate. Recurrence was defined as the reappearance of disease after a complete response. Patients who experienced death without local failure, biochemical failure prior to local failure, and development of distant metastases prior to local failure were censored on the date of the competing event. The corresponding outcome time was measured from the date of randomization. Due to an insufficient number of events (2 in each arm), this endpoint was not statistically compared. Local control rates at 4 years were calculated using the Kaplan-Meier method.
Time Frame: From randomization to date of local failure, death, or last follow-up. Analysis occurs after all patients have been potentially followed for 4 years.
Population: Eligible patients who did not withdraw consent
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Androgen Suppression + Radiation Therapy | Androgen Suppression + Radiation Therapy + Chemotherapy
Number analyzed (Participants) | 281 | 282
percentage of participants | 99.2 [97.0 to 99.8] | 99.5 [96.6 to 99.9]

4. Secondary Outcome: Distant Metastasis
Description: Distant failure was considered when there was evidence of metastatic disease. Patients who experienced death without distant failure, local failure prior to distant failure, and biochemical failure prior to distant failure were censored on the date of the competing event. The corresponding outcome time was measured from the date of randomization. Distant failure rates at 4 year were calculated using the Kaplan-Meier method.
Time Frame: From randomization to date of distant metastasis, death, or last follow-up. Analysis occurs after all patients have been potentially followed for 4 years.
Population: Eligible patients who did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Androgen Suppression + Radiation Therapy | Androgen Suppression + Radiation Therapy + Chemotherapy
Number analyzed (Participants) | 281 | 282
percentage of participants | 2.6 [1.1 to 5] | 1.9 [0.7 to 4.1]
Statistical Analysis 1: Comparison: Androgen Suppression + Radiation Therapy vs Androgen Suppression + Radiation Therapy + Chemotherapy; Distant failure rates at 4 years were calculated using the Kaplan-Meier method and compared by a two-side log-rank test at the 0.05 significance level; Test type: Superiority or Other; p = 0.21, Log Rank

5. Secondary Outcome: Disease-free Survival
Description: A failure for disease-free survival is the first of the following: biochemical failure, local failure, distant metastases, or death due to any cause. The corresponding outcome time was measured from the date of randomization. Disease-free survival rates at 4 years were calculated using the Kaplan-Meier method.
Time Frame: From randomization to date of progression, death, or last follow-up. Analysis occurs after all patients have been potentially followed for 4 years.
Population: Eligible patients who did not withdraw consent.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Androgen Suppression + Radiation Therapy | Androgen Suppression + Radiation Therapy + Chemotherapy
Number analyzed (Participants) | 281 | 282
percentage of participants | 73.0 [67.4 to 77.9] | 78.5 [73.1 to 82.9]
Statistical Analysis 1: Comparison: Androgen Suppression + Radiation Therapy vs Androgen Suppression + Radiation Therapy + Chemotherapy; Disease-free survival rates were compared by a two-sided log-rank test at a significance level of 0.05; Test type: Superiority or Other; p = 0.0484, Log Rank

6. Secondary Outcome: Incidence of Adverse Events
Description: Adverse events are graded using CTCAE v3.0. The worst grade of all adverse events for each patient is counted.
Time Frame: From start of treatment until the end of follow-up
Population: Eligible patients who started protocol treatment and did not withdraw consent
Measure: Number; unit: percentage of participants
Arm/Group | Androgen Suppression + Radiation Therapy | Androgen Suppression + Radiation Therapy + Chemotherapy
Number analyzed (Participants) | 281 | 282
percentage of participants
  Grade 1 | 14.9 | 2.1
  Grade 2 | 48.4 | 25.9
  Grade 3 | 26.0 | 40.1
  Grade 4 | 4.3 | 28.4
  Grade 5 | 1.4 | 0.7

7. Secondary Outcome: The Time Interval Between Biochemical Failure and Distant Failure Respect to Testosterone Level
Description: Biochemical failure is defined as the first of either prostate-specific antigen (PSA) failure or the initiation of salvage hormone therapy. PSA failure is defined as a rise in PSA of 2 ng/ml over the nadir PSA. Distant failure is defined as the first occurrence of distant metastasis.
Time Frame: From date of biochemical failure to development of distant metastasis. Maximum follow-up was 12.9 years.
Population: The analysis will not be done because testosterone measurement dates were not collected.
Arm/Group | Androgen Suppression + Radiation Therapy | Androgen Suppression + Radiation Therapy + Chemotherapy
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Validity of PSA Endpoint as a Surrogate for Overall Survival
Description: Prentice's operational criteria for determining whether determining whether biochemical failure (surrogate endpoint) is a suitable endpoint for overall survival (true endpoint):
  1. Treatment is prognostic for true endpoint
  2. Treatment is prognostic for surrogate endpoint
  3. Surrogate is prognostic for true endpoint
  4. The full effect of the treatment on the true endpoint is explained by the surrogate.
  If any of the criteria are not met, it is concluded that biochemical failure is not a suitable surrogate for overall survival. Therefore, if any of the criteria are met, the other criteria do not do not need to be evaluated.
Time Frame: From randomization to last follow-up. Analysis occurs after all patients have been potentially followed for 4 years.
Population: Because the second criterion is not met, further analysis was not performed.
Arm/Group | Androgen Suppression + Radiation Therapy | Androgen Suppression + Radiation Therapy + Chemotherapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Participants who started protocol treatment.
Arm/Group | Androgen Suppression + Radiation Therapy | Androgen Suppression + Radiation Therapy + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 26/302 | 93/302
Other Adverse Events (participants affected / at risk) | 278/302 | 289/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Androgen Suppression + Radiation Therapy (N=302) | Androgen Suppression + Radiation Therapy + Chemotherapy (N=302)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 12
Hemoglobin (Blood and lymphatic system disorders) | 0 | 10
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 3
Cardiac general - Other (Cardiac disorders) | 1 | 3
Myocardial ischemia (Cardiac disorders) | 6 | 5
Myocarditis NOS (Cardiac disorders) | 0 | 1
Ventricular arrhythmia NOS (Cardiac disorders) | 0 | 2
Abdominal pain NOS (Gastrointestinal disorders) | 0 | 2
Colitis NOS (Gastrointestinal disorders) | 0 | 2
Colonic hemorrhage (Gastrointestinal disorders) | 0 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Diarrhea NOS (Gastrointestinal disorders) | 1 | 9
Gastritis NOS (Gastrointestinal disorders) | 0 | 1
Gastrointestinal - Other (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Pancreatitis NOS (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting NOS (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 1 | 0
Edema: limb (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 4
Multi-organ failure (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Sudden death (General disorders) | 3 | 0
Syndromes - Other (General disorders) | 0 | 1
Hypersensitivity NOS (Immune system disorders) | 0 | 1
Bladder infection NOS (Infections and infestations) | 0 | 1
Infection - Other (Infections and infestations) | 1 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Brain + Spinal cord (encephalomyelitis) (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils: Blood (Infections and infestations) | 0 | 1
Infection with unknown ANC: Skin (cellulitis) (Infections and infestations) | 0 | 1
Kidney infection NOS (Infections and infestations) | 1 | 0
Lymph gland infection (Infections and infestations) | 0 | 1
Pneumonia NOS (Infections and infestations) | 1 | 0
Urinary tract infection NOS (Infections and infestations) | 1 | 1
Dermatitis radiation NOS (Injury, poisoning and procedural complications) | 1 | 0
Fracture NOS (Injury, poisoning and procedural complications) | 1 | 1
Vascular access NOS complication (Injury, poisoning and procedural complications) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 2
Hypercholesterolemia (Investigations) | 1 | 1
Leukopenia NOS (Investigations) | 0 | 24
Lymphopenia (Investigations) | 0 | 4
Metabolic/laboratory - Other (Investigations) | 1 | 1
Neutrophil count (Investigations) | 0 | 34
Platelet count decreased (Investigations) | 1 | 1
Troponin I increased (Investigations) | 0 | 2
Weight decreased (Investigations) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 4
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 2
Hyperglycemia NOS (Metabolism and nutrition disorders) | 0 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal/soft tissue - Other (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Secondary Malignancy - possibly related to cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cerebral ischemia (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1
Neurology - Other (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 1
Euphoric mood (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Libido decreased (Psychiatric disorders) | 0 | 1
Cystitis NOS (Renal and urinary disorders) | 1 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 3
Renal failure NOS (Renal and urinary disorders) | 1 | 3
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1
Ejaculatory disorder NOS (Reproductive system and breast disorders) | 0 | 1
Erectile dysfunction NOS (Reproductive system and breast disorders) | 0 | 4
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary/upper respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatology/skin - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Localised exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Sweating increased (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flushes NOS (Vascular disorders) | 2 | 2
Hypertension NOS (Vascular disorders) | 0 | 1
Hypotension NOS (Vascular disorders) | 1 | 2
Peripheral ischemia (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Androgen Suppression + Radiation Therapy (N=302) | Androgen Suppression + Radiation Therapy + Chemotherapy (N=302)
Blood/bone marrow - Other (Blood and lymphatic system disorders) | 3 | 18
Hemoglobin (Blood and lymphatic system disorders) | 37 | 176
Lacrimation increased (Eye disorders) | 2 | 16
Abdominal pain NOS (Gastrointestinal disorders) | 15 | 23
Constipation (Gastrointestinal disorders) | 29 | 54
Diarrhea NOS (Gastrointestinal disorders) | 153 | 159
Dyspepsia (Gastrointestinal disorders) | 6 | 25
Fecal incontinence (Gastrointestinal disorders) | 16 | 13
Gastrointestinal - Other (Gastrointestinal disorders) | 20 | 25
Hemorrhoids (Gastrointestinal disorders) | 15 | 13
Nausea (Gastrointestinal disorders) | 13 | 81
Proctitis NOS (Gastrointestinal disorders) | 43 | 47
Rectal hemorrhage (Gastrointestinal disorders) | 37 | 41
Stomatitis (Gastrointestinal disorders) | 0 | 29
Vomiting NOS (Gastrointestinal disorders) | 8 | 18
Edema: limb (General disorders) | 15 | 51
Fatigue (General disorders) | 157 | 235
Pain - Other (General disorders) | 16 | 26
Alanine aminotransferase increased (Investigations) | 16 | 31
Aspartate aminotransferase increased (Investigations) | 17 | 23
Blood alkaline phosphatase increased (Investigations) | 7 | 15
Leukopenia NOS (Investigations) | 20 | 145
Lymphopenia (Investigations) | 24 | 63
Metabolic/laboratory - Other (Investigations) | 4 | 25
Neutrophil count (Investigations) | 3 | 107
Platelet count decreased (Investigations) | 11 | 34
Weight decreased (Investigations) | 6 | 17
Weight increased (Investigations) | 21 | 40
Anorexia (Metabolism and nutrition disorders) | 7 | 33
Hyperglycemia NOS (Metabolism and nutrition disorders) | 16 | 103
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 32
Hypokalemia (Metabolism and nutrition disorders) | 2 | 16
Hyponatremia (Metabolism and nutrition disorders) | 3 | 28
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 64
Back pain (Musculoskeletal and connective tissue disorders) | 25 | 43
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 18
Muscle weakness NOS (Musculoskeletal and connective tissue disorders) | 16 | 23
Musculoskeletal/soft tissue - Other (Musculoskeletal and connective tissue disorders) | 7 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 36
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 29
Dizziness (Nervous system disorders) | 8 | 29
Dysgeusia (Nervous system disorders) | 2 | 53
Peripheral motor neuropathy (Nervous system disorders) | 6 | 19
Peripheral sensory neuropathy (Nervous system disorders) | 20 | 110
Anxiety (Psychiatric disorders) | 7 | 15
Depression (Psychiatric disorders) | 20 | 20
Insomnia (Psychiatric disorders) | 22 | 53
Libido decreased (Psychiatric disorders) | 65 | 63
Bladder pain (Renal and urinary disorders) | 6 | 18
Cystitis NOS (Renal and urinary disorders) | 33 | 46
Pollakiuria (Renal and urinary disorders) | 209 | 210
Renal/genitourinary - Other (Renal and urinary disorders) | 39 | 47
Urinary incontinence (Renal and urinary disorders) | 34 | 47
Urinary retention (Renal and urinary disorders) | 55 | 56
Urogenital hemorrhage (Renal and urinary disorders) | 10 | 15
Ejaculatory disorder NOS (Reproductive system and breast disorders) | 22 | 24
Erectile dysfunction NOS (Reproductive system and breast disorders) | 122 | 120
Gynecomastia (Reproductive system and breast disorders) | 20 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 41
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 27 | 68
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 119
Dermatitis exfoliative NOS (Skin and subcutaneous tissue disorders) | 7 | 28
Dermatology/skin - Other (Skin and subcutaneous tissue disorders) | 13 | 24
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 18
Nail disorder NOS (Skin and subcutaneous tissue disorders) | 1 | 51
Sweating increased (Skin and subcutaneous tissue disorders) | 14 | 22
Hot flushes NOS (Vascular disorders) | 206 | 192
Hypertension NOS (Vascular disorders) | 8 | 15

LIMITATIONS AND CAVEATS:
Due to insufficient number of events, local control analysis was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.